CLINICAL TRIAL: NCT02201823
Title: A PHASE I/Ib, FIRST IN HUMAN, DOSE-ESCALATION STUDY OF ABTL0812 IN PATIENTS WITH ADVANCED SOLID TUMOURS
Brief Title: Phase I/Ib Clinical Trial of ABTL0812 in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ability Pharmaceuticals SL (Industry)
Collaborators: Hospital Clinic of Barcelona (Other); Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-C1-2013; 2013-001293-17 (EudraCT Number); PEI 13-057 (Other: AEMPS)
Record Dates: First submitted 2014-05-09; First posted 2014-07-28 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — ABTL0812

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABTL0812 (Experimental): ABTL0812 oral
  Interventions: Drug: ABTL0812

INTERVENTIONS:
Drug: ABTL0812 — ABTL0812. Five cohorts and one extension phase.

SUMMARY:
Ability Pharmaceuticals promotes a clinical trial to determine the adequate dose of a new drug, ABTL0812, that will be administered orally daily to patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase I/Ib, unicenter, open-label and single-agent study. This study consists of two different parts, a dose escalation phase and an extension phase in patients with advanced solid tumors.

ABTL0812 will be administered orally, daily, for 28 days (considered cycle 1). First endpoint is to determine the Maximum Tolerated Dose (MTD). MTD is defined as the highest dose at which no more than one in six patients experiences a ABTL0812 related Dose-Limiting Toxicity (DLT). DLT will be evaluated during the first treatment cycle.

Dose escalation phase will be performed with an accelerated design of 3 + 3

Once the 28 days cycle has finished, patients may continue receiving ABTL0812 on a daily continuous schedule if the patient is deemed to have clinical benefit from treatment, according to the treating physician. Treatment will continue until disease progression, onset of unacceptable drug toxicities, or patient/physician's request to discontinue.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Willing and able to provide informed consent
* Patients with histologically or cytologically confirmed diagnosis of advanced solid tumour refractory to standard treatment or for whom no effective therapy exists
* Evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* All female subjects will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically Female subjects of childbearing potential must agree to use two forms of highly effective contraception methods during the study and for a period of 6 months following the last administration of the study drug. Male subjects and their female partners who are of childbearing potential and are not practicing total abstinence, must agree to use two forms of highly effective contraception during the study and for a period of 6 months following the last administration of the study drug
* Adequate bone marrow function
* Adequate coagulation profile
* Adequate hepatic function
* Adequate renal function
* Life expectancy of at least 3 months, in the opinion of the investigator
* Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ grade 1 (as defined by Common Terminology Criteria for Adverse Events version 4.02).
* Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol

Exclusion Criteria:

* Patients receiving treatment within 4 weeks prior to study entry with an investigational drug, chemotherapy, targeting agents or hormonal therapy (patients may continue to receive Luteinizing-hormone-releasing hormone analogue therapy for prostate cancer in face of rising PSA), radiation (except to bone) or surgery (except exploratory biopsy or intravenous device implantation, etc.) (6 weeks for nitrosoureas or Mitomycin C, or for investigational drug within 5 half-lives of the treatment, whichever is longer). Participation in non-interventional or observational studies is allowed.
* Patients with symptomatic brain metastases. Patients with asymptomatic brain metastases can be included in the study if they are kept on stable doses of steroids for a period of 1 month prior to study entry.
* Patients with gastrointestinal abnormalities including inability to take oral medications, malabsorption syndromes or other clinically significant gastrointestinal abnormalities that may impair the absorption of the investigational medicinal product.
* Pregnancy or lactation. Serum pregnancy test to be performed within 7 days prior to study treatment start.
* Patients with myocardial infarction within ≤ 12 months prior to study entry, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina pectoris, or unstable cardiac arrhythmia requiring medication.
* Evidence of preexisting uncontrolled hypertension. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Patients with known Hepatitis B or C or human immunodeficiency virus (HIV) infection
* Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that in the opinion of the investigator may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of ABTL0812, administered orally on a daily continuous schedule in adult patients with advanced solid tumours | First 28 days of treatment

SECONDARY OUTCOMES:
To assess safety and tolerability of ABTL0812 | First 28 days of treatment
To evaluate preliminary antitumour activity of ABTL0812 | After 6 months of treatment
To determine the recommended Phase II dose | First 28 days of treatment

OTHER OUTCOMES:
To evaluate the pharmacokinetic (PK) profile of ABTL0812 in patients with advanced solid tumours | First 28 days of treatment
To evaluate the pharmacodynamic (PD) profile of ABTL0812 exploring preliminary biomarkers of drug activity | First 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vidal, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Polonio-Alcala E, Sole-Sanchez S, Munoz-Guardiola P, Megias-Roda E, Perez-Montoyo H, Yeste-Velasco M, Alfon J, Lizcano JM, Domenech C, Ruiz-Martinez S, Puig T. ABTL0812 enhances antitumor effect of paclitaxel and reverts chemoresistance in triple-negative breast cancer models. Cancer Commun (Lond). 2022 Jun;42(6):567-571. doi: 10.1002/cac2.12282. Epub 2022 Mar 16. No abstract available. PMID 35293148
- [Derived] Vidal L, Victoria I, Gaba L, Martin MG, Brunet M, Colom H, Cortal M, Gomez-Ferreria M, Yeste-Velasco M, Perez A, Rodon J, Sohal DPS, Lizcano JM, Domenech C, Alfon J, Gascon P. A first-in-human phase I/Ib dose-escalation clinical trial of the autophagy inducer ABTL0812 in patients with advanced solid tumours. Eur J Cancer. 2021 Mar;146:87-94. doi: 10.1016/j.ejca.2020.12.019. Epub 2021 Feb 12. PMID 33588149